CLINICAL TRIAL: NCT05654753
Title: RANDOMIZED DOUBLE BLIND CONTROLLED STUDY ASSESSING THE EFFICACY OF FECAL MICROBIOTA TRANSPLANTATION IN PATIENTS WITH AXIAL SPONDYLOARTHRITIS RESISTANT TO CONVENTIONAL TREATMENT
Brief Title: The Efficacy of Fecal Microbiota Transplatation on Axial Spondyloarthritis Patients Resistant to Conventional Treatment
Acronym: FMT-SpA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Arthritis & Clarins Worldwide 2016 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP220934; 2023-504852-89-00 (Registry Identifier: Eu CT Number)
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Axial Spondyloarthritis
Keywords: Axial Spondyloarthritis; dysbiotic microbiota; Fecal microbiota transplantation; eubiotic microbiota
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): active FMT
  Interventions: Drug: active FMT
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: active FMT — MaaT033®, a lyophilized full-ecosystem intestinal microbiota delayed release oral capsule containing native, donor-derived (pooled from 4-6 donors) microbiome product manufactured by MaaT Pharma® will be delivered orally. Patients will receive 20 Maat033 capsules, each containing approximatively 0.42 g of microbiome product at once at day 0, then 3 capsules/day from day 1 through day 20.
  Arms: Experimental
Drug: Placebo — Patients will receive 20 capsules placebo, each containing placebo at once at day 0, then 3 capsules/day from day 1 through day 20.
  Arms: Placebo

SUMMARY:
Current pharmacological management of inflammatory rheumatism and in particular axial SpA remains imperfect. Only 50% of patients respond to the most effective biotherapies, and many of them are only partially relieved. In addition, these are extremely expensive treatments that expose them to the risk of potentially serious side effects. Compelling evidence indicates that gut dybiosis could be a critical trigger of inflammation in axial SpA and thus correcting dysbiosis represents an attractive way of reversing the pathogenic process.The efficacy of FMT in patients with axial SpA has never been studied. This randomized double-blind study will be the first to assess feasability of FMT in axial SpA, the capacity of this procedure to restore healthy microbiome, its tolerance and its potential efficacy on disease activity. If sucessfull, this trial would set the path to larger-scale clinical trials of FMT to treat axial SpA.

Two-co primary objectives in a hierarchical design:

* to evaluate the capacity of FMT to correct dysbiosis in active axial SpA despite well-conducted phamacological treatment by replacing pre-existing dysbiotic microbiota with healthier microbiota.
* to explore the efficacy of FMT versus placebo on clinical evolution of SpA.

DETAILED DESCRIPTION:
Axial spondyloarthritis (SpA) is a chronic inflammatory disease primarily affecting the sacroiliac and spinal joints that usually begins in young adults and is a major cause of chronic pain and disability that profoundly alter the quality of life of patients. Besides non-steroidal anti-inflammatory drugs, the development of anti-tumor necrosis factor-α (TNFα) and anti-interleukin (IL-17) biotherapies and of JAK inhibitors, has improved the management of these patients. However only half of the patients respond to these treatments and many of them are only partially relieved. Remarkably, this disorder frequently combines with overt inflammatory bowel disease (IBD) -i.e. Crohn's disease (CD) or ulcerative colitis (UC)- and even more frequently with subclinical gut inflammation, leading to suspect a role of the gut microbiota as a possible trigger. Consistently, recent studies evidenced an alteration of gut microbiota composition -or dysbiosis- in the course of SpA that appeared all the more pronounced that disease was more active. It was notably shown a restriction of bacterial diversity and an expansion of species considered as potentially pro-inflammatory, including Ruminococcus gnavus. Given its potential involvement in the pathogenesis of SpA, gut microbiota could be considéred as a promising therapeutic target. Fecal microbiota transplantation (FMT) is a technic consisting in thorough replacement of dysbiotic microbiota by healthy dondor's microbiota that has recently been developped to correct dysbiosis. It has been validated for the treatment of intractable colitis due to Clostridium difficile and its efficacy has been reported in CD or UC. The current trial, aims to evaluate efficacy of FMT in drug-resistant axial SpA.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age 18 to 75 years old) with SpA, meeting the ASAS classification criteria for axial SpA, with presence of radiographic sacro-illitis (ankylosing spondylitis) or not.
* Patient suffering of active SpA, with or without treatment, having a BASDAI score ≥ 4 (0-10) at baseline and a score of back pain ≥ 4 (0-10) despite optimal drug management for at least 6 months including at least 2 different NSAIDs at the maximum tolerated dose for at least 2 months (or less in case of intolerance or contra-indication) and at least a first line of biotherapy (anti-TNFα or anti-IL-17) for at least 4 months (or less in case of intolerance or contra-indication).
* Subjects are allowed to continue NSAID, sulfasalazin (≤ 3 g/day) and/or methotrextae ( ≤ 25 mg/week) and/or hydroxychloroquine (≤ 400 mg/day) and/or oral corticosteroid (≤ 10 mg/day of prednisone), as long as these treatments have remained at stable dose for 4 weeks prior to baseline.
* Subjects are allowed to continue anti-TNFα, anti-IL-17 or JAKinhibitor therapies, as long as these treatments have remained at stable dose for 3 months prior to baseline.
* Women of childbearing potential with efficient contraceptive protection at the inclusion and during at least the interventional phase (D168).
* Patient with health insurance (AME except).
* Patient is willing to provide written informed consent prior to enrolment and agrees to follow the protocol.

Exclusion Criteria:

1. Patient under legal protection (guardianship or curatorship)
2. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development
3. Pregnant or breastfeeding woman
4. Patient with IBD in active state, according to the judgment of the Investigator
5. Corticosteroid injection within 4 weeks before inclusion
6. Active infection according to the judgment of the Investigator
7. Any antibiotic (including Sulfasalazin) or antifungal treatment within 4 weeks before inclusion
8. Probiotics intake within 4 weeks before inclusion
9. Known infection with Clostridoides difficile or Escherichia coli within 10 days before inclusion
10. Patients with unstable severe condition other than axial SpA on that could jeopardize treatment procedure or evaluation according to the investigator's assessment
11. Previous FMT treatment
12. Contra-indication to colon preparation (Moviprep® or Moviprep orange®) according to SmPC
13. Current or past evidence of bowel obstruction
14. Confirmed or suspected intestinal ischemia
15. Confirmed or suspected toxic megacolon or gastrointestinal perforation
16. Extended colectomy (> two-thirds of colon)
17. Any gastro-intestinal bleeding in the past 3 months before inclusion
18. Any history of gastro-intestinal surgery in the past 3 months before inclusion
19. Severe organ dysfunction
20. Any contra-indication to swallow capsules
21. Known allergy or intolerance to IMP and / or excipients according to Investigator's Brochure
22. Lack of access to a refrigerator to store the medication (MaaT033® or MaaT030®)
23. Concomitant participation in another interventional clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Increase in gut Metagenome Species Pangenome (MSP) richness in the "intervention" arm. | at baseline and D 42
  Fecal microbiota composition will be assessed by thorough microbial DNA sequencing (shotgun) at baseline (anytime between D-4 and D-1) and then at D28, D42, D84 and D168. The success will be evaluated by an increase in gut Metagenome Species Pangenome (MSP) richness over the period of study.
The proportion of patients satisfying ASAS 20 improvement criteria by randomization group | at D 42
  ASAS20 is defined by an improvement of ≥ 20% and of ≥ 10 points on a 0-100 numerical scale of 3 of the 4 following domains: global evaluation by the patient (PGA), pain, Bath Ankylosing Spondylitis Functional Index (BASFI) and inflammation (evaluated by the answer to both last questions of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)) as well as an absence of deterioration from baseline by ≥ 20% and by ≥ 10 points in the fourth domain. The comparison of ASAS20 scores at D42 between randomization groups will be an exploratory analysis, considering literature data.

SECONDARY OUTCOMES:
efficacy of FMT | week 6
  Superior efficacy of FMT over placebo defined by an increase in MSP richness at week 6 in the FMT group, superior to variation in the placebo group
Change of dysbiotic fecal microbiota | at baseline, at weeks 3, 12 and 24
  To correct dysbiotic fecal microbiota at weeks 3, 12 and 24 in FMT-treated group, by comparison with baseline. Fecal microbiota composition will be assessed by thorough microbial DNA sequencing (shotgun), in a way similar to week 6 in FMT and placebo groups and the variation between baseline and different end-points (weeks 3, 12, 24) will be compared between both arms.
Clinical improvement | at baseline, weeks 3, 6, 12 and 24
  Clinical improvement during the 24 weeks follow-up after FMT or sham-FMT. We will compare between both arms the proportion of patients satisfying ASAS20 improvement criteria at weeks 3, 6, 12 and 24 as compared to baseline (week 0).
  [ASAS20 is defined by an improvement of at least 20% and of at least 10 points on a 0-100 scale in ≥ 3 of the following 4 domains: global assessment by the patient (PGA), back pain, Bath Ankylosing Spondylitis Functional Index (BASFI) and inflammation (evaluated by the answer to both last questions of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) and absence of deterioration in the potential remaing domain, where deterioration is defined as a change for the worse of ≥ 20% and net worsening of ≥ 10 points (on a scale of 0-100)
ESR and CRP levels | at weeks 3, 6, 12 and 24
  Improvement of biological inflammation by ESR and CRP levels variation
CHANGE OF ASDAS_CRP and ASDAS_ESR | at weeks 3, 6, 12 and 24
  Improvement of ASDAS_CRP and ASDAS_ESR at weeks 3, 6, 12 and 24
Change in Bath Ankylosing Spondylitis Metrology Index | at weeks 3, 6, 12 and 24
  Improvement of Bath Ankylosing Spondylitis Metrology Index (BASMI) at weeks 3, 6, 12 and 24
non-steroidal anti-inflammatory drugs (NSAID) intake | through study completion, an average of 18 months
  Decrease of non-steroidal anti-inflammatory drugs (NSAID) intake score.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Breban, MD, PhD, Principal Investigator — Rheumatology Department - Ambroise Paré hospital - APHP
Locations (1):
- Rheumatology Department, Ambroise Paré hospital - APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No